CLINICAL TRIAL: NCT05943977
Title: A Randomized, Open Label, 2-Period, Cross-over Study to Evaluate the Bioequivalence of the Oversea Manufactured Sample and Domestic Manufactured Sample in Single Intravenous Dose of MB-102 (Relmapirazin) (Part I), and an Efficacy Study to Assess the Performance of the MediBeacon Transdermal GFR Measurement System and Domestic Manufactured Sample of MB-102 (Relmapirazin) for Evaluation of Kidney Function in Chinese Normal and Renal Compromised Subjects (Part II)
Brief Title: A Bioequivalence and Efficacy Study of MB-102 (Relmapirazin) in Chinese Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Collaborators: MediBeacon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HDNP102-301; CTR20230300 (Registry Identifier: www.chinadrugtrials.org.cn)
Record Dates: First submitted 2023-03-22; First posted 2023-07-13 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Kidney Diseases; Kidney Injury; Kidney Failure
Keywords: Glomerular Filtration Rate; Relmapirazin; Pharmacokinetics; MB-102
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency | interventions — relmapirazin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- 130 mg MB-102 DMID, then 130 mg MB 102-OMID (Experimental): Participants will receive a single 130 mg dose of the MB-102 Domestic Manufactured Investigational Drug (DMID), and blood and urine samples will be collected per protocol. There will be a 5-day washout period between treatments, and then participants will receive a single 130 mg dose of the MB-102 Overseas Manufactured Investigational Drug (OMID). Blood and urine samples will be collected per protocol
  Interventions: Drug: MB-102 DMID; Drug: MB-102 OMID
- 130 mg MB-102 OMID, then 130 mg MB 102-DMID (Experimental): Participants will receive a single 130 mg dose of the MB-102 Overseas Manufactured Investigational Drug (OMID), and blood and urine samples will be collected per protocol. There will be a 5-day washout period between treatments, and then participants will receive a single 130 mg dose of the MB-102 Domestic Manufactured Investigational Drug (DMID). Blood and urine samples will be collected per protocol.
  Interventions: Drug: MB-102 DMID; Drug: MB-102 OMID
- Participants with eGFR ≥ 70 mL/min/1.73 m^2 (Experimental): 130 mg of the MB-102 Domestic Manufactured Investigational Drug (DMID) will be administered to participants with estimated glomerular filtration rate (eGFR) eGFR ≥ 70 mL/min/1.73 m^2, and fluorescence measured using the MediBeacon Transdermal GFR Measurement System
  Interventions: Drug: MB-102 DMID; Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (TGFR)
- Participants with eGFR < 70 mL/min/1.73 m^2 (Experimental): 130 mg of the MB-102 Domestic Manufactured Investigational Drug (DMID)will be administered to participants with estimated glomerular filtration rate (eGFR) eGFR < 70 mL/min/1.73 m^2, and fluorescence measured using the MediBeacon Transdermal GFR Measurement System
  Interventions: Drug: MB-102 DMID; Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (TGFR)

INTERVENTIONS:
Drug: MB-102 DMID — 130 mg of the MB-102 Domestic Manufactured Investigational Drug administered by intravenous injection over 30-60 seconds, followed by a 10 mL normal saline flush administered over 30-60 seconds.
  Other Names: Relmapirazin
Drug: MB-102 OMID — 130 mg of the MB-102 Overseas Manufactured Investigational Drug (OMID) administered by intravenous injection over 30-60 seconds, followed by a 10 mL normal saline flush administered over 30-60 seconds.
  Other Names: Relmapirazin
  Arms: 130 mg MB-102 DMID, then 130 mg MB 102-OMID; 130 mg MB-102 OMID, then 130 mg MB 102-DMID
Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (TGFR) — On treatment day, participants will have the TGFR sensor placed on their chests, and the MediBeacon Transdermal GFR Measurement System will be initiated to collect background fluorescence. When this is completed, participants will then receive a single dose of MB-102. Fluorescent measurements terminated by the system when a low signal-to-noise threshold is reached.
  Arms: Participants with eGFR < 70 mL/min/1.73 m^2; Participants with eGFR ≥ 70 mL/min/1.73 m^2

SUMMARY:
Part I (bioequivalence) will evaluate the bioequivalence of the Oversea Manufactured Sample (used in the MediBeacon Phase 3 Study 100-103; NCT05425719) and Domestic Manufactured Sample in Single Intravenous Dose of MB-102 (Relmapirazin) in healthy Chinese adults. Part II (efficacy) will evaluate the performance of the MediBeacon Transdermal GFR Measurement System and Domestic Manufactured Sample of MB-102 (Relmapirazin) for Evaluation of Kidney Function in Chinese participants.

DETAILED DESCRIPTION:
Part I (bioequivalence) will be conducted as an open-label, 2-period, 2-treatment, crossover study with 24 subjects expected to enroll. Blood and urine samples will be collected. Part II (efficacy) will enroll up to 100 subjects, divided into 2 strata (1:1) in accordance with screening eGFR measured by the CKD-EPI equation. Blood samples will be collected at predefined time points and the MediBeacon Transdermal GFR Measurement System will be used to collect fluorescent measurements.

ELIGIBILITY:
Inclusion Criteria:

Bioequivalence study:

1. The participant is aged 18-55 years, inclusive, at the date of informed consent

   1. Eligible female non-pregnant participants who are either not of child-bearing potential or willing to use adequate contraception during the trial and at least 1 month post-dose
   2. Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 1 month post-dose
   3. For women of child-bearing potential, the participant should have a negative serum pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly during the trial and at least 1 month post-dose, i.e. abstinence, oral contraceptive either combined or progesterone alone; injectable progesterone, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, IUD device or system or male partner sterilization
2. The participant weighs at least 50 kg, and has a body mass index (BMI) between 19 and 25 kg/m2, inclusive, at Screening
3. The participant is a Chinese healthy adult male or female
4. Men will not donate sperm during the study and for 1 month following the last dose of study drug
5. Participants who are capable of directly providing informed consent and who can comply with the requirements and restrictions required by the protocol
6. Adequate venous access sufficient to allow blood sampling per protocol requirements

Efficacy study:

1. Age > 18 years - male or female

   1. Eligible female non-pregnant participants who are either not of child-bearing potential or willing to use adequate contraception during the trial and at least 1 month post-dose
   2. Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 1 month post-dose
   3. For women of child-bearing potential, the participant should have a negative serum pregnancy test at Screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly during the trial and at least 1 month post-dose, i.e. abstinence, oral contraceptive either combined or progesterone alone; injectable progesterone, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, IUD device or system or male partner sterilization
   4. Men will not donate sperm during the study and for 1 month following the last dose of study drug
2. Participants who are capable of directly providing informed consent and who can comply with the requirements and restrictions required by the protocol
3. Adequate venous access sufficient to allow blood sampling per protocol requirements

Exclusion Criteria:

Bioequivalence study:

1. Participants positive via PCR testing for COVID-19
2. Recent donation or loss of blood or plasma: 100 mL to 499 mL within 30 days prior to the initial dose of the study medication; or more than 499 mL within 56 days prior to the initial dose of study medication
3. Non-steroidal anti-inflammatory (NSAID) use within 3 days of MB-102 dosing.
4. The participant has participated in a clinical trial and has received an investigational product within the following time ranges: prior to the first dosing day in the current study: either 30 days or 5 half-lives of the investigational product (whichever duration is longer).
5. History of severe allergic hypersensitivity reactions (unacceptable adverse events) or anaphylactoid reaction to any allergen including drugs, MB-102 or other related products (intolerance to a drug is not considered a drug allergy).
6. Participants with positive serum pregnancy test
7. The participant has an abnormal (clinically significant) electrocardiogram (ECG) at Screening or prior to the study drug administration in Period 1
8. The participant has abnormal laboratory values that suggest a clinically significant underlying disease, or subject with the following abnormalities at Screening or prior to the study drug administration in Period 1: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 x the upper limits of normal (ULN)
9. History of drug and/or alcohol abuse within the past year.
10. Participants with a creatine kinase (CK) value of greater than the upper limit of normal that is not explainable by exercise and that does not come back to reference range upon retest;
11. Any reason which, in the opinion of the Principal Investigator or Medical Sub-Investigator, would prevent the participant from safely participating in the study.

Efficacy study:

1. Participants positive via PCR testing for COVID-19
2. Recent donation or loss of blood or plasma: 100 mL to 499 mL within 30 days prior to the initial dose of the study medication; or more than 499 mL within 56 days prior to the initial dose of study medicatio
3. Non-steroidal anti-inflammatory (NSAID) use within 3days of MB-102 dosing.
4. The participant has participated in a clinical trial and has received an investigational product within the following time ranges: prior to the first dosing day in the current study: either 30 days or 5 half-lives of the investigational product (whichever duration is longer).
5. History of skin sensitivity to adhesives (e.g. Band-Aids, surgical tape)
6. History of severe allergic hypersensitivity reactions (unacceptable adverse events) or anaphylactoid reaction to any allergen including drugs, MB-102 or other related products (intolerance to a drug is not considered a drug allergy).
7. Any characteristics such as acute or chronic medical condition or cardiac or laboratory or physical examination abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of the study results in the judgement of the investigator and would make the subject inappropriate for entry into this study.
8. Significant scarring, tattoos or alterations in pigmentation on the sternum or other sensor location testing areas that would alter sensor readings versus other areas of the skin
9. Use of tanning sprays, tanning products etc. on the upper chest within 2 weeks of dosing day; Use of makeup, lotions, Vaseline or other products on the area of the upper chest on the day prior to or the day of dosing
10. Any serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, or psychiatric condition that in the opinion of the investigator would limit the participants' ability to complete study requirements or may put the participant at increased risk or compromise the interpretability of study results.
11. Currently receiving dialysis
12. Currently anuric
13. Participants with positive serum pregnancy test
14. Participants with an eGFR >120 mL/min/1.73m2 or <15 mL/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of MB-102 | Pre-dose (within 60 minutes prior to dosing) and at 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes (±2 minutes), 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 20 hours and 24 hours (±5 minutes) post-dose
  Blood samples will be collected pre-dose (within 60 minutes prior to dosing) and at 5 min, 15 min, 30 min, 60 min, 90 min (±2 min), 2h, 3h, 4h, 5h, 6h, 8h, 10h , 12h, 16h, 20h and 24h (±5 min) post-dose, and will be analyzed using validated analytical methods. The area under the plasma concentration-time curve (ng*hr/mL) from time 0 to infinity will be calculated as: AUC0-last+Clast//λz where Clast is the predicted concentration (based on the terminal regression) at the time of the last measurable concentration.
Correlation of transdermal derived glomerular filtration rate (tGFR) to the plasma-derived indexed glomerular filtration rate (nGFR) | Up to 24 hours
  Statistical agreement between tGFR and nGFR will be calculated using P30 statistics

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of MB-102 | Pre-dose (within 60 minutes prior to dosing) and at 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes (±2 minutes), 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 20 hours and 24 hours (±5 minutes) post-dose
  Blood samples will be collected pre-dose (within 60 minutes prior to dosing) and at 5 min, 15 min, 30 min, 60 min, 90 min (±2 min), 2h, 3h, 4h, 5h, 6h, 8h, 10h , 12h, 16h, 20h and 24h (±5 min) post-dose, and will be analyzed using validated analytical methods.Maximum plasma concentration (Cmax; measured in ng/mL) will be directly determined from the concentration-time data.
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration for MB-102 (AUC0-last) | Pre-dose (within 60 minutes prior to dosing) and at 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes (±2 minutes), 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 20 hours and 24 hours (±5 minutes) post-dose
  Blood samples will be collected pre-dose (within 60 minutes prior to dosing) and at 5 min, 15 min, 30 min, 60 min, 90 min (±2 min), 2h, 3h, 4h, 5h, 6h, 8h, 10h , 12h, 16h, 20h and 24h (±5 min) post-dose, and will be analyzed using validated analytical methods.The area under the plasma concentration-time curve (ng*hr/mL) will be estimated from time 0 to the last measurable concentration using noncompartmental analyses.
The terminal rate constant (Lambda_z) of MB-102 | Pre-dose (within 60 minutes prior to dosing) and at 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes (±2 minutes), 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 20 hours and 24 hours (±5 minutes) post-dose
  Blood samples will be collected pre-dose (within 60 minutes prior to dosing) and at 5 min, 15 min, 30 min, 60 min, 90 min (±2 min), 2h, 3h, 4h, 5h, 6h, 8h, 10h , 12h, 16h, 20h and 24h (±5 min) post-dose, and will be analyzed using validated analytical methods. The terminal rate constant (λz) will be determined by linear regression of the terminal linear phase of the log plasma concentration-time profile.
Total plasma clearance (CL) of MB-102 | Pre-dose (within 60 minutes prior to dosing) and at 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes (±2 minutes), 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 20 hours and 24 hours (±5 minutes) post-dose
  Blood samples will be collected pre-dose (within 60 minutes prior to dosing) and at 5 min, 15 min, 30 min, 60 min, 90 min (±2 min), 2h, 3h, 4h, 5h, 6h, 8h, 10h , 12h, 16h, 20h and 24h (±5 min) post-dose, and will be analyzed using validated analytical methods. Total plasma clearance (the volume of plasma cleared of the drug over time) will be calculated as: Clp = Dose/ AUC0-inf.
Volume of distribution (Vd) of MB-102 | Pre-dose (within 60 minutes prior to dosing) and at 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes (±2 minutes), 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 20 hours and 24 hours (±5 minutes) post-dose
  Blood samples will be collected pre-dose (within 60 minutes prior to dosing) and at 5 min, 15 min, 30 min, 60 min, 90 min (±2 min), 2h, 3h, 4h, 5h, 6h, 8h, 10h , 12h, 16h, 20h and 24h (±5 min) post-dose, and will be analyzed using validated analytical methods. Volume of distribution will be calculated by Vd=CL/λz
The elimination half-life of MB-102 | Pre-dose (within 60 minutes prior to dosing) and at 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes (±2 minutes), 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 20 hours and 24 hours (±5 minutes) post-dose
  Blood samples will be collected pre-dose (within 60 minutes prior to dosing) and at 5 min, 15 min, 30 min, 60 min, 90 min (±2 min), 2h, 3h, 4h, 5h, 6h, 8h, 10h , 12h, 16h, 20h and 24h (±5 min) post-dose, and will be analyzed using validated analytical methods.The elimination half-life (the time required for the concentration of the drug to reach half of its original value) will be calculated as t1/2 λz= ln(2)/ λz.
Time to Maximum Plasma Concentration (Tmax) of MB-102 | Pre-dose (within 60 minutes prior to dosing) and at 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes (±2 minutes), 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 20 hours and 24 hours (±5 minutes) post-dose
  Blood samples will be collected pre-dose (within 60 minutes prior to dosing) and at 5 min, 15 min, 30 min, 60 min, 90 min (±2 min), 2h, 3h, 4h, 5h, 6h, 8h, 10h , 12h, 16h, 20h and 24h (±5 min) post-dose, and will be analyzed using validated analytical methods.The time to maximum plasma concentration (Tmax; measured in minutes) will be directly determined from the concentration-time data.
Area under the plasma concentration-time curve extrapolated as a percentage of the total (AUC_%Extrap) | Pre-dose (within 60 minutes prior to dosing) and at 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes (±2 minutes), 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 20 hours and 24 hours (±5 minutes) post-dose
  Blood samples will be collected pre-dose (within 60 minutes prior to dosing) and at 5 min, 15 min, 30 min, 60 min, 90 min (±2 min), 2h, 3h, 4h, 5h, 6h, 8h, 10h , 12h, 16h, 20h and 24h (±5 min) post-dose, and will be analyzed using validated analytical methods. AUC_%Extrap will be calculated as (AUC0-inf-AUC0-last)/AUC0-inf *100%.
Number of participants with treatment-emergent adverse events associated with the MediBeacon Transdermal GFR Measurement System device | Up to 10 days
  An adverse event is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, temporally associated with the use of a medicinal product, whether or not related to the investigational medical device or drug

CONTACTS AND LOCATIONS:
Overall Officials: Yuanyuan Luo, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Dong Sun, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Yanxia Yu, Principal Investigator — Suzhou Municipal Hospital
Locations (2):
- China (2):
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Affiliated hospital of Xuzhou Medical University, Xuzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No